CLINICAL TRIAL: NCT07161609
Title: The Effect of Different Types of Masks on Surgical Smoke Exposure
Brief Title: The Effect of Masks on Surgical Smoke Exposure
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Seher Gürdil Yılmaz, PhD , Department of Surgical Nursing, Principal investigator, Asst. Prof., Mersin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Different Types of Masks
Record Dates: First submitted 2025-09-05; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Surgical Smoke
Keywords: Surgical smoke; Particle; Mask; Operating room team

STUDY DESIGN:
Intervention Model Description: Prospective, parallel, three-arm, randomized controlled clinical trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: When the researchers (E.D., S.Ü., and S.GY.) enter the operating room, they will open the numbered envelope provided by the coordinating researcher (G.A.U.) to determine the group assignment of the surgery. All researchers other than the coordinating researcher will be blinded to the group allocations. The study data will be entered into a computer by another researcher (C.K.), who is not involved in the data collection process, in order to ensure blinding during data analysis and reporting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single surgical mask (Experimental): During the surgery of patients undergoing hip prosthesis, an air sample will be collected to determine the particle count by attaching a single surgical mask to the tip of the particle counter.
  Interventions: Device: Particle counter
- Double surgical mask (Experimental): During the surgery of patients undergoing hip prosthesis, an air sample will be collected to determine the particle count by attaching a double surgical mask to the tip of the particle counter.
  Interventions: Device: Particle counter
- N95 mask (Experimental): During the surgery of patients undergoing hip prosthesis, an air sample will be collected to determine the particle count by attaching a N95 surgical mask to the tip of the particle counter.
  Interventions: Device: Particle counter

INTERVENTIONS:
Device: Particle counter — The collection of air samples will begin with the surgical incision and will continue for 10 minute

SUMMARY:
Surgical smoke refers to the gaseous plume released into the air as a result of the thermal destruction of tissues by energy-based devices used in operating rooms. The composition of surgical smoke may include various organic compounds. In the literature, the most frequently identified chemical substances in surgical smoke are formaldehyde, acrolein, hydrocarbons, fatty acids, hydrocyanic acid, phenols, nitriles, acrylonitrile, hydrogen cyanide, benzene, and toluene. These particles can negatively affect the health of the operating room personnel. According to current guidelines, masks are recommended as the primary personal protective equipment to prevent respiratory exposure associated with surgical smoke. During surgical procedures, operating room staff frequently use surgical masks. Although surgical masks are the most commonly preferred personal protective equipment to protect healthcare workers against microorganisms and aerosols, they are unfortunately ineffective in filtering small particles. Therefore, the present study aimed to determine the impact of different types of masks on exposure to surgical smoke.

DETAILED DESCRIPTION:
With the advancement of surgical techniques, the instruments and devices used in surgery have also rapidly evolved. Among these are energy-based devices that produce heat to achieve dissection or hemostasis during surgical procedures. Surgical smoke refers to the gaseous plume released into the air as a result of the thermal destruction of tissues by such devices, and is also termed cautery smoke, smoke plume, aerosol, or bioaerosol. While approximately 95% of surgical smoke consists of water vapor, the remaining 5% contains dead and viable cellular material, blood particles, viruses, bacteria, and toxic gases. The quantity and particle size of surgical smoke vary depending on factors such as the type of energy source, the tissue treated, and the duration and extent of treatment.

Surgical smoke has been identified by professional associations as a chemical hazard affecting the safety of operating room environments. Larger particles (≥5 μm) deposit in the nasal and oropharyngeal regions, particles of 2-5 μm can reach the airways, and particles <2 μm may penetrate lung tissue, accumulating in bronchioles and alveoli. Various toxic chemicals have been identified in surgical smoke, including formaldehyde, acrolein, hydrocarbons, fatty acids, hydrogen cyanide, phenols, nitriles, acrylonitrile, benzene, and toluene. Studies have also reported the presence of volatile organic compounds such as toluene, xylene, ethylbenzene, styrene, and naphthalene, with concentrations varying by procedure type.

Exposure to surgical smoke negatively impacts the health of operating room staff, with reported symptoms such as headaches, nausea, throat irritation, cough, eye problems, respiratory difficulties, dermatitis, and anxiety. To mitigate these risks, recommended measures include staff education, awareness programs, installation of smoke evacuation systems, use of personal protective equipment, and development of institutional protocols.

Among personal protective equipment, masks are the primary barrier recommended against respiratory exposure to surgical smoke. Although surgical masks are widely used to protect healthcare professionals against microorganisms and aerosols, they are largely ineffective in filtering fine particles. Professional guidelines advise the use of N95 respirators in conjunction with smoke evacuation systems, especially in procedures with high risk of viral transmission, given their superior filtration capacity.

However, studies specifically examining the effectiveness of different types of masks against surgical smoke remain limited, with most research focusing on mask performance during the COVID-19 pandemic. Experimental studies comparing filtration efficiency have demonstrated superior performance of N95/FFP2 respirators compared to surgical masks. In this context, the present study aims to investigate the effectiveness of different mask types in protecting operating room staff from surgical smoke exposure.

ELIGIBILITY:
Inclusion Criteria:

* Use of electrocautery,
* Duration of surgery longer than 2 hours,
* Elective total or partial hip prosthesis procedures.

Exclusion Criteria:

* No use of electrocautery,
* Duration of surgery shorter than 2 hours,
* Emergency total or partial hip prosthesis procedures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in airborne particle count | The number of particles in the air collected during the 10 minutes following the initiation of the surgical incision.
  Difference in particle count between masks

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
In order to avoid duplication, it is not intended to be shared until the research is completed.

REFERENCES:
- [Background] Dikmen Aydın, Y., Gürkan, A., & Kırtıl, İ. (2024). Cerrahi duman: Ameliyathanede çalışan sağlık profesyonellerine etkisi ve alınan önlemlerin incelenmesi. Sağlık ve Yaşam Bilimleri Dergisi, 6(1), 40-47.